CLINICAL TRIAL: NCT04031209
Title: Retrospective and Prospective Multi-Center Outcomes Study of G7 Dual Mobility System Used in Total Hip Arthroplasty for the Treatment of Femoral Neck Fracture
Brief Title: G7 Dual Mobility System Used in Total Hip Arthroplasty for the Treatment of Femoral Neck Fracture
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CSA2019-02H
Record Dates: First submitted 2019-07-04; First posted 2019-07-24 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- G7 G7 Acetabular System: All patients will receive G7 G7 Acetabular System
  Interventions: Device: G7 Acetabular System

INTERVENTIONS:
Device: G7 Acetabular System — All patients will receive G7 Acetabular System

SUMMARY:
This is a retrospective and prospective, multi-center, non-comparative, post market clinical follow-up study involving orthopedic surgeons skilled in THA and experienced implanting the devices included in this study.

DETAILED DESCRIPTION:
The objectives of the study are to document the performance and safety of the G7 Dual Mobility System when used in primary total hip arthroplasty for the treatment of femoral neck fracture by analysis of standard scoring systems, radiographs, revision and adverse event records.The study will include a maximum of 15 centers and up to 300 implanted hips. Each center may enroll up to a maximum of 40 hips to permit the consistency of outcomes across a variety of investigators and clinical setting

ELIGIBILITY:
Inclusion Criteria:

* 55 to 80 years of age, inclusive
* Skeletally mature
* Have undergo treatment or in need of primary THA treatment of non-union, femoral neck fracture, unmanageable by other techniques
* Have G7 Dual Mobility system implanted or decision to have a G7 Dual Mobility system implanted was made independently and prior to recruitment into study
* Willing and able to complete scheduled follow-up evaluations as described in the study protocol
* Has participated in the Informed Consent process and is willing and able to sign an IRB/EC approved informed consent

Exclusion Criteria:

* Is septic, has an active infection or has osteomyelitis at the affected joint
* Has significant osteoporosis as defined by treating surgeon
* Has metabolic disorder(s) which may impair bone formation
* Has osteomalacia
* Has distant foci of infections which may spread to the implant site
* Has rapid joint destruction, marked bone loss or bone resorption on pre-operative radiographs
* Has vascular insufficiency, muscular atrophy at the implant site or neuromuscular disease which might jeopardize the outcome of the surgery
* Has any concomitant disease which is likely to jeopardize the functioning or success of the implant
* Is known to be pregnant
* Is a prisoner, known alcohol or drug abuser or mentally incompetent or unable to understand what participation in this study entails
* Has a known sensitively or allergy to one or more of

Ages: 55 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients who required primary THA for treatment of femoral neck fracture and satisfy eligibility criteria outlined in this section. In order to avoid potential selection bias, each investigator will offer study participation to each consecutive eligible patient presenting as a candidate for primary THA using G7 Dual Mobility System.
Sampling Method: Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Implant dislocation rate | One year post-surgery
  Dislocation is defined as the complete loss of articulation contact between two artificial joint components.

SECONDARY OUTCOMES:
Pain and Functional Performance by Oxford Hip Score | Up to 5 years post-surgery
  The Oxford Hip score consist of 12 disease-specific questions measuring patient-reported pain and function of the hip joint. Responses to each question are formatted as a 5-point Likert scale, scored from 0 (the worst outcome/most symptoms) to 4 (the best outcome / least symptoms). The scores for each question are added together for a final result between 0 and 48.
Implant survivorship by revision rates | Up to 5 years post-surgery
  Cumulative survival rates using a Kaplan-Meier analysis.
Quality of life by EQ-5D-5L questionnaire | Up to 5 years post-surgery
  This 5-level EQ-5D version (EQ-5D-5L) consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. A 1-digit number expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The health states may be converted into a single index value where 1 represents full health and 0 represents death. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Quality of life by JHEQ | Up to 5 years post-surgery
  The Japanese Orthopaedic Association hip disease evaluation questionnaire (JHEQ) is a self-administered questionnaire that evaluates the quality of life in patients with hip disease. The questionnaire consists of three subscales: pain (28 points), movement (28 points), and mental (28 points), with higher scores indicating a better outcome. This measurement is applicable to Japanese population only.
Pain and Functional Performance by JOA Hip Score | Up to 5 years post-surgery
  The Japanese Orthopaedic Association (JOA) hip score consists of four subcategories: pain (Pain, 40 points), range of motion (ROM, 20 points), ability to walk (Gait, 20 points), and activities of daily life (ADL, 20 points), with higher scores indicating a better outcome. This measurement is applicable to Japanese population only.
Adverse events reported | Up to 5 years post-surgery
  Summary of adverse events by category, incidence and frequency

CONTACTS AND LOCATIONS:
Overall Officials: Kee-Hyung Rhyu, Principal Investigator — Kyunghee University Medical Center
Locations (7):
- South Korea (7):
  - Seoul National University Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Asan medical Centre, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - KyungHee University Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No